CLINICAL TRIAL: NCT02126098
Title: Cohort Study of Chinese Patients With Pulmonary Vasculitis
Brief Title: Observation Study of Clinical Manifestation and Outcome in Chinese Patients With Pulmonary Vasculitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-PULMONARY DISEASES; 2011BA11B17 (Other Grant/Funding Number: 2011BA11B17the Ministry of Science and Technology of China)
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: ANCA-associated Vasculitis; Granulomatosis With Polyangiitis; Microscopic Polyangiitis; EosinphilicGranulomatosis With Polyangiitis
Keywords: ANCA-associated vasculitis; Granulomatosis with polyangiitis; Microscopic polyangiitis; Wegner's granulomatosis; Eosinphilic granulomatosis with polyangiitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Biospecimen Retention: Samples With DNA — serum lymphocytes urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adults who diagosed ANCA-vasculitis: Patients with Wegener's granulomatosis or microscopic polyangiitis were eligible to participate in the study if they had
  1. Positive serum assays for proteinase 3-ANCA or myeloperoxidase-ANCA
  2. manifestations of severe disease,11 and a Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) of 3 or more (scores range from 0 to 63, with higher scores indicating more active disease)

SUMMARY:
The purpose of this study is to observe the clinical manifestation, Lab findings including chest CT scans, pathological findings and outcomes in chinese patients with pulminary vasculitis.

DETAILED DESCRIPTION:
Presentation of patient with suspected vasculitis

1. Established diagnosis Clinical findings Laboratory workup Tissue biopsy Angiogram where appropriate
2. Evaluating respiratory system Chest HRCT Pulmonary function test Bronchoscopy exam(BALF, TBB) Lung biopsy(needle biopsy, VAST)
3. screening underlying damage to other system Paranasal sinus, vision & audition Nervous system Kidney Gastrointestinal tract Heart & vessel Skin Hematology Muscle, bone & joint
4. Treatment
5. Prognosis

Evaluation

1. Study visits occurred at baseline; at weeks 4; and at 2, 4, 6,12,18,24,30 months.
2. Disease activity was measured on the basis of the BVAS/WG and the physician's global assessment.
3. Damage related to disease or treatment was scored according to the Vasculitis Damage Index (scores for this index range from 0 to 64, with higher scores in- dicating more severe damage).
4. Health related quality of life was scored with the use of the Med- ical Outcomes Study 36-Item Short-Form Health Survey (SF-36).Scores on this scale range from 0 to 100, with higher scores indicating better health.
5. Serial serum samples were tested for proteinase 3-ANCA and myeloperoxidase-ANCA by means of a direct enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Aged from 18-75 years with informed consent
* Patients with ANCA-vasculitis

  1. Wegener's granulomatosis, microscopic polyangiitis or CSS
  2. positive serum assays for proteinase 3-ANCA or myeloperoxidase-ANCA
  3. manifestations of activity disease, and Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) of 3 or more (scores range from 0 to 63, with higher scores indicating more active disease)

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Secondary vasculitis, cancer,infective disease or drug induced vasculitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who newly diagnosed ANCA-vasculitis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Completely Remission | 6 months
  BVAS/WG of 0 and successful completion of the prednisone taper at 6 months.

SECONDARY OUTCOMES:
Disease flare | during the period of observation(30months)
  Disease flare
  1. an increase in the BVAS/WG of 1 point or more.
  2. Patients were classified as having early treatment failure if at 1 month their BVAS/WG had not decreased by at least 1 point or a new manifestation of disease had emerged.

OTHER OUTCOMES:
Adverse events | during the period of observation (30months)
  1. deaths (from all causes)
  2. malignant conditions
  3. grade 2 or higher leukopenia or thrombocytopenia
  4. grade 3 or higher infections
  5. drug induced cystitis
  6. venous thromboembolic events
  7. stroke
  8. hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Juhong Shi, M.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China